CLINICAL TRIAL: NCT00938743
Title: Driving Ability in Adults With ADHD Before and After 10-weeks of Treatment With 40-80mg Atomoxetine vs. Untreated Adults With ADHD
Brief Title: Driving in Adults With Attention-deficit/Hyperactivity Disorder (ADHD) Before and During Treatment With Atomoxetine
Acronym: DrivPerfATX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Esther Sobanski, MD, Central Institute of Mental Health, Mannheim
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007-004309-90
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2011-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; adults; driving performance; atomoxetine
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atomoxetine (Active Comparator): Treatment with a final dosis of 40-80mg atomoxetine daily
  Interventions: Drug: Atomoxetine
- Waiting list (No Intervention)

INTERVENTIONS:
Drug: Atomoxetine — 40-80 mg atomoxetine once daily, including titration 10 weeks
  Arms: Atomoxetine

SUMMARY:
According available data individuals with ADHD are impaired in their driving ability which can be improved by stimulant medication. The impact of the specific noradrenalin-reuptake-inhibitor atomoxetine on driving ability of patients with ADHD has never been studied so far.

The present study aims to evaluate the effects of atomoxetine treatment in patients with ADHD on practical driving abilities which will be assessed with a standardized driving test, a structured one-week driving diary and driving related neuropsychological processing especially different aspects of attention and executive functions which will be assessed with a neuropsychological test battery designed for the assessment of drivers fitness. A functional magnetic resonance imaging (fMRI) - investigation will also be performed at the beginning and after a 10-week treatment with atomoxetine. The study will be conducted in a single-blind placebo controlled parallel group design in cooperation of the academic Adult ADHD-outpatient clinics of the Central Institute of Mental Health, Mannheim and the Institute of Legal and Traffic Medicine of the University of Heidelberg, Germany.

It is expected that treatment with atomoxetine will improve practical driving abilities and driving related neuropsychological processing. It is expected that risk taking and impulsive decision making will be reduced and sustained attention and overview of complex traffic situations will be improved while driving.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent Form signed by the patients.
2. Patients are 16-50 years of age when the informed consent document is obtained (Visit 1).
3. Patients have been judged by the investigator to be reliable to keep appointments for clinic visits and all tests, including venipuncture and examinations, required by the protocol.
4. Patients must meet DSM-IV-TR criteria for ADHD assessed by the Conners' Adult ADHD Diagnostic Interview for DSM-IV (CAADID) and KIDDIE-SADDS-PL respectively and according to expert consensus.
5. Patients must also have a significant other evaluation of their current ADHD using the Conners' Adult ADHD Rating Scale Observer: Screening Version (CAARS-O: SV) and Conners' Rating Scales- Revised (CRS-R):SV respectively
6. Patients must have a CGI-ADHD-S score of more than 4 points (moderate symptoms) at Visit 1.
7. Patients aged 18 and older must have a valid driver's license.
8. Patients must have laboratory results assessed at Visit 1, including serum chemistries, haematology, and thyroid function, that show no significant abnormalities. Significant would include laboratory deviations requiring acute medical intervention or further medical evaluation.
9. Patients must have a negative urinary drug screen at Visit 1.
10. Patients must have no medical history of heart disease that could be destabilized by increases in heart rate or blood pressure. The screening electrocardiogram (ECG) performed at Visit 1 must not show significant abnormalities. Significant would include a heart rate of less than 40 bpm and more than 120 bpm respectively, any disturbances in rhythm and conduction as well as ECG-findings pointing to myocardial infarction.
11. Females of childbearing potential defined as women not surgically sterilized and between menarche and 1 year post-menopause must test negative for pregnancy at Visit 1 based on an urinary pregnancy test and agree to use a reliable method of birth control (e.g., oral contraceptives, a reliable barrier method of birth control like diaphragms, intrauterine devices; partner with vasectomy or abstinence) during the study.

Exclusion Criteria:

* The exclusion criteria are designed to eliminate patients who do not meet study population criteria or whose participation in the study would be inappropriate due to underlying safety issues and to ensure that patients participating in the study are in a stable physical condition. They further are designed to maintain consistency with the approved global labeling for atomoxetine.

Patients will be excluded from the study if they meet any of the following criteria:

1. Patients who are investigator site personnel directly affiliated with the study, or are immediate family of investigator site personnel directly affiliated with the study. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
2. Patients who meet full DSM-IV diagnostic criteria for any history of bipolar or psychotic disorder, current major depression, current generalized anxiety disorder or panic disorder will be excluded from the study. Assessment will be done by clinical history and a Structured Clinical Interview for DSM-IV Axis-I disorders (SCID).
3. Patients who are currently using alcohol, drugs of abuse, or any prescribed or over-the-counter medication in a manner which the investigator considers indicative of abuse or who meet DSM-IV-TR criteria for substance abuse, assessed by clinical history and a Structured Clinical Interview for DSM-IV (SCID). Patients must not use drugs of abuse or illicitly obtained prescription drugs during the study, and a urine drug screen may be obtained at any time during the study. Alcohol use should be discouraged, and if, in the investigator's judgment, the patient is using alcohol to excess, the patient should be discontinued.
4. Patients, who in the opinion of the investigator, are at serious suicidal or homicidal risk.
5. Patients with organic brain disease, for example, dementia, traumatic brain injury residual, or a history of any seizure disorder (except febrile seizures during childhood).
6. Patients with a history of severe allergies to more than one class of medications or multiple adverse drug reactions.
7. Patients who have a known history of narrow angle glaucoma.
8. Males with prostatic symptoms.
9. Patients with significant medical conditions that are likely to become unstable during the trial or would likely be destabilized by treatment with atomoxetine, (for example, cardiovascular disease that would be at aggravated by increased heart-rate), or require treatment with excluded medications.
10. Patients who have any medical condition or who are taking a medication on a daily basis (for example albuterol, inhalation aerosols) that has sympathomimetic activity.
11. Patients with hypertension. For the purposes of this protocol, hypertension will be defined as average systolic or diastolic blood pressure, measured on at least 2 separate occasions, greater than or equal to 140/90. Patients whose blood pressure is controlled with non-excluded medication are eligible for inclusion.
12. Patient taking any psychotropic medications on a daily basis within 2 weeks before Visit1. However, zolpidem to a dose of 10 mg may be used intermittently as needed for insomnia provided they are not used more than 3 times weekly.
13. Patients who have received regular treatment within the last 30 days with a drug that has not received regulatory approval for any indication or taking any antipsychotic medication at the time of study entry.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Standardized practical driving test | 1/2010

SECONDARY OUTCOMES:
Action-Reaction-Test Battery | 1/2010
Performance criteria for drivers' fitness according to the "Guidelines of Driver Fitness" | 1/2010
Safety measures including vital signs, laboratory test, ECG, assessment of SAEs | 1/2010

CONTACTS AND LOCATIONS:
Locations (1):
- Central Institute of Mental Health, Adult ADHD Outpatient Department, Mannheim, Germany